CLINICAL TRIAL: NCT06461520
Title: Effects of Maze Balance Board Training Program on Balance in Children With Hearing Impairment.
Brief Title: Effects of Maze Balance Board Training on Balance in Children With Hearing Impairment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0785
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hearing Impaired Children
Keywords: Hearing Loss; Balance; Pediatric balance scale; Maze balance board training; SWOC test
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: It will be a Randomized Controlled Trial in which non-convenient probability sampling will be used. Two groups of 5-8 yrs age will be formed in which participants will be randomly divided. Group A will undergo maze balance board training for 60 minutes a day twice a week. Group B will undergo proprioceptive training of 40 minutes thrice a week
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask both groups about treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maze Balance Board (Experimental): Every child will have their balance evaluated using the SWOC tool, CTSIB, and Pediatric Balance Scale. Patients performed a range of proprioceptive exercises, such as static one-leg standing, board balancing, squatting, and 20 minutes of straight-line walking on a hard surface before moving to a foam surface. For 20 minutes each session, proprioceptive exercises were conducted with open eyes first, followed by closed ones. The training program for the maze balancing board will next take place. There will be seven phases to the maze balance board training; each stage will last for two days and there will be three sessions per day, each lasting an hour.
  Interventions: Other: Maze Balance board; Other: Proprioceptive training
- Proprioceptive training (Active Comparator): This group will get proprioceptive training. For a total of ten weeks, the intervention will be carried out three times a week for forty minutes each. Without maze-balance board training, the training schedule will consist of three sessions each week, lasting ten minutes each for preparatory, twenty minutes for proprioceptive, and ten minutes for restorative activities. Every meeting ended with a 10-minute cool-down and 10-minute warm-up to signify the quality of work.
  Interventions: Other: Proprioceptive training

INTERVENTIONS:
Other: Maze Balance board — Every child will have their balance evaluated using the SWOC tool, CTSIB, and Pediatric Balance Scale. Patients performed a range of proprioceptive exercises, such as static one-leg standing, board balancing, squatting, and 20 minutes of straight-line walking on a hard surface before moving to a foam surface. For 20 minutes each session, proprioceptive exercises were conducted with open eyes first, followed by closed ones. The training program for the maze balancing board will next take place. There will be seven phases to the maze balance board training; each stage will last for two days and there will be three sessions per day, each lasting an hour.
  Arms: Maze Balance Board
Other: Proprioceptive training — This group will get proprioceptive training. For a total of ten weeks, the intervention will be carried out three times a week for forty minutes each. Without maze-balance board training, the training schedule will consist of three sessions each week, lasting ten minutes each for preparatory, twenty minutes for proprioceptive, and ten minutes for restorative activities. Every meeting ended with a 10-minute cool-down and 10-minute warm-up to signify the quality of work.

SUMMARY:
The majority of children's everyday activities need balance, which is the complex ability to maintain, obtain, or restore the condition of balance of the body when a child is standing still, getting ready to move, or getting ready to stop moving. Integration of several sensory, motor, and biomechanical inputs is necessary for balance. Nonetheless, alterations in certain sensory systems (such as visual, somatosensory, and vestibular) may result in imbalances inside the body. Previous research has demonstrated that children and adolescents with hearing impairments are more likely to experience balance and/or motor deficits as a result of vestibular system damage, which increases their risk of developing motor and balance issues. Additionally, research has demonstrated a link between hearing loss and a higher risk of all-cause death, maybe through physical activity-related factors including balance and mobility. Combining maze control training with traditional physical therapy's proprioceptive exercises tests your balance and improves your stability overall.

DETAILED DESCRIPTION:
Balance is the complex ability to retain, achieve, or restore the condition of equilibrium of the body whether a kid is standing still, getting ready to move, or getting ready to stop moving. It is necessary for most of the everyday activities that children engage in. Balance requires the integration of multiple sensory, motor, and biomechanical inputs. However, changes in some sensory systems (visual, somatosensory, vestibular) might lead to internal disequilibrium. Previous studies have shown that vestibular system damage in children and adolescents with hearing impairments increases the likelihood of balance and/or motor deficiencies, which in turn raises the chance of developing motor and balance difficulties. Furthermore, studies have shown a connection between hearing loss and an increased risk of dying from all causes, maybe as a result of elements connected to physical activity, such as mobility and balance. By combining proprioceptive exercises from standard physical therapy with maze control training, you may test your balance and enhance your general stability.

For this, a randomized controlled trial will be employed. The study will be approved by the ethics committee. when that, patients who fulfill the study's inclusion requirements will be included when their informed consent has been obtained. The 36 patients will be divided into two groups, and each child's balance will be assessed using the pediatric balance scale, CTSIB, and SWOC. The control group will participate in a regular 10-week physical therapy program that includes 60 minutes of proprioceptive training for balance two times a week, while the study group will receive the proprioceptive training along-with seven-stage maze balance board training three times per day and twice a week for a total of 60 minutes. The data will be examined for mean and standard deviation using SPSS 25. A suitable assessment will be employed to contrast the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Children of age 5-8yrs with moderate to severe hearing impairment (41-80 decibels )
* Ability to understand the command
* Single leg stance (Screening Test): Putting leg down before 30 sec using arm for balance
* No history of MSK disorder.

Exclusion Criteria:

* Children with perceptual or visual deficits
* Children with seizures or epilepsy
* Marked hip and knee flexion contractures
* Serious medical complications
* Children with fixed deformity of both lower limbs and children with surgical interventions, e.g., tendon release

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-06-16 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | Baseline and 8 weeks
  A modified version of the Berg Balance Scale which is known as the Pediatric Balance Scale is used to evaluate children's functional balance abilities. The 14 items on the scale have a maximum score of 56 points and are rated from 0 (lowest function) to 4 (highest function). It has good inter-rater reliability (ICC=0.997) and test-retest reliability (ICC=0.098). The pediatric balance scale's validity (r=0.797, p <0.05)
Standardized Walking Obstacle Course (SWOC) | Baseline and 8 weeks
  Physical therapists can evaluate a patient's mobility, balance, coordination and functional ability to navigate obstacles using a standardized walking obstacle course tool. The aim is to replicate actual circumstances and obstacles that people might face in their day-to-day pursuits.
  For both time and step count, the inter-rater reliability of the SWOC scores was also determined to be extremely high. It was found that for both time and step count, the intra-rater (test-retest) reliability of the SWOC was extremely or very highly reliable. The concurrent validity of the SWOC was investigated by looking at correlations between time and step count on both the TUG and SWOC conditions. With p-values less than 0.003, all Pearson product-moment correlation coefficients were judged significantly.
Modified Clinical Test of Sensory Interaction in Balance (CTSIB TEST): | Baseline and 8 weeks
  The test is a therapist's adaptation of the Computerized Dynamic Posturography, which measures our ability to maintain our balance in the face of gravity by means of our visual, vestibular, and somatosensory interactions. Shumway-Cook and Horak created the exam in 1986, and in 1987, it was further explored as a potential clinical tool. It has been demonstrated that manipulating visual and support surface information causes difficulties for patients with uncompensated unilateral vestibular impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Wardah Haroon, MS*, Principal Investigator — Riphah International University Lahore
Locations (1):
- Children Hospital Faislabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis A, Hind S. The impact of hearing impairment: a global health problem. Int J Pediatr Otorhinolaryngol. 1999 Oct 5;49 Suppl 1:S51-4. doi: 10.1016/s0165-5876(99)00213-x. PMID 10577775
- [Background] Emmett SD, West KP Jr. Nutrition and hearing loss: a neglected cause and global health burden. Am J Clin Nutr. 2015 Nov;102(5):987-8. doi: 10.3945/ajcn.115.122598. Epub 2015 Oct 14. No abstract available. PMID 26468119
- [Background] Jafari Z, Kolb BE, Mohajerani MH. Age-related hearing loss and tinnitus, dementia risk, and auditory amplification outcomes. Ageing Res Rev. 2019 Dec;56:100963. doi: 10.1016/j.arr.2019.100963. Epub 2019 Sep 23. PMID 31557539